CLINICAL TRIAL: NCT05226845
Title: Is Patient Choice of Exercise Preference Important in Chronic Neck Pain? A Randomized Clinical Study
Brief Title: Is Patient Choice of Exercise Preference Important in Chronic Neck Pain?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Alexander Achalandabaso, Principal Investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Alcalá University
Record Dates: First submitted 2021-12-04; First posted 2022-02-07 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Chronic Neck Pain
Keywords: Chronic neck pain; Physical Exercise; Kinesiophobia; Cervical strength; Adherence to treatment
MeSH Terms: conditions — Motor Activity; Kinesiophobia; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise to improve the neck strength in neck pain chosen by the therapist (Experimental)
  Interventions: Other: prescribed exercise
- exercise to improve the neck strength in neck pain chosen by the patient (Experimental)
  Interventions: Other: chosen exercise

INTERVENTIONS:
Other: prescribed exercise — the therapist chooses the five exercises to do
  Arms: exercise to improve the neck strength in neck pain chosen by the therapist
Other: chosen exercise — the patient chooses the five exercises to perform among fifteen possibilities
  Arms: exercise to improve the neck strength in neck pain chosen by the patient

SUMMARY:
Nonspecific chronic neck pain is the third most frequent problem in Spain. It has an annual presence between 15% and 50% where women are the most affected. This pain influences the psychosocial state of the person. Physical exercise has been shown to be effective in a wide variety of chronic pain conditions, including improving quality of life and emotional problems. Design: Single-blind, controlled, randomized clinical trial. Methods: The study will be approached in the Faculty of Nursing and Physiotherapy of the University of Alcalá. 52 subjects with nonspecific chronic neck pain will be selected and randomly divided into two groups. The first group should perform 5 exercises that have been shown to be effective in the management of neck pain selected by the physiotherapist focused on neck pain. The second group must choose, from a list of exercises that have been shown to be effective in the management of neck pain, 5 exercises. Both groups should record the pain, the number of repetitions and the series performed. The duration of the intervention will be a total of 8 weeks with evaluations pre-intervention, post-intervention and 4 weeks after the end of the intervention. The objective of this study is to evaluate if the exercise chosen by the patient is better than the exercises selected by the physiotherapist for the variables chronic neck pain, strength of the affected muscles, kinesiophobia and adherence to treatment.

ELIGIBILITY:
Inclusion Criteria:

* chronic neck pain

Exclusion Criteria:

* Spine surgery, shoulder girdle or cervical area surgery, whether traumatic or not.
* Rheumatic pathology.
* Impaired cognitive function.
* Vascular pathology that prevents exercise.
* Cardiopulmonary pathology that prevents exercise.
* Fear of any of the tests or measurements to be carried out.
* Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Changes in Disability | Baseline, 8 weeks (primary timepoint) and 4 weeks after intervention.
  using the Neck Disability Index Questionnaire. It is a scale whose values range from 0 to 50. The higher the score, the greater the disability.

SECONDARY OUTCOMES:
Changes in kinesiophobia | Baseline, 8 weeks (primary timepoint) and 4 weeks after intervention.
  using Tampa scale of kinesiophobia (TSK-11). It is a scale whose values range from11 to 44. The higher the score, the greater the kinesiophobia.
Changes in muscular endurance | Baseline, 8 weeks (primary timepoint) and 4 weeks after intervention.
  using Grimmer test
Adherence to treatment | Baseline, 8 weeks (primary timepoint) and 4 weeks after intervention.
  using a journal entry
changes in pain | Baseline, 8 weeks (primary timepoint) and 4 weeks after intervention.
  Using the visual analog scale. It is a 100-mm long horizontal line. Zero means no pain, 100-mm means the worst pain imaginable.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Alexander achalandabaso, Alcalá de Henares, Madrid
  - Universidad de Alcalá, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geneen LJ, Moore RA, Clarke C, Martin D, Colvin LA, Smith BH. Physical activity and exercise for chronic pain in adults: an overview of Cochrane Reviews. Cochrane Database Syst Rev. 2017 Apr 24;4(4):CD011279. doi: 10.1002/14651858.CD011279.pub3. PMID 28436583
- [Background] Ambrose KR, Golightly YM. Physical exercise as non-pharmacological treatment of chronic pain: Why and when. Best Pract Res Clin Rheumatol. 2015 Feb;29(1):120-30. doi: 10.1016/j.berh.2015.04.022. Epub 2015 May 23. PMID 26267006
- [Background] Polaski AM, Phelps AL, Kostek MC, Szucs KA, Kolber BJ. Exercise-induced hypoalgesia: A meta-analysis of exercise dosing for the treatment of chronic pain. PLoS One. 2019 Jan 9;14(1):e0210418. doi: 10.1371/journal.pone.0210418. eCollection 2019. PMID 30625201
- [Background] Sluka KA, Frey-Law L, Hoeger Bement M. Exercise-induced pain and analgesia? Underlying mechanisms and clinical translation. Pain. 2018 Sep;159 Suppl 1(Suppl 1):S91-S97. doi: 10.1097/j.pain.0000000000001235. PMID 30113953